CLINICAL TRIAL: NCT00513474
Title: Rasburicase to Prevent Graft -Versus-Host Disease
Brief Title: Rasburicase in Preventing Graft-Versus-Host Disease in Patients With Hematologic Cancer or Other Disease Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Bimalangshu Dey, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000558480; MGH-07-071; DFCI-07-071
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: graft versus host disease; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; Waldenström macroglobulinemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; previously treated myelodysplastic syndromes; primary myelofibrosis; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic eosinophilic leukemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; refractory hairy cell leukemia; refractory multiple myeloma; secondary acute myeloid leukemia; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Hairy Cell | interventions — Busulfan; Cyclophosphamide; Cyclosporins; Etoposide; Methotrexate; rasburicase; Sirolimus; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; fludarabine; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasburicase Group (Experimental): Myeloablative (bone marrow depletion) conditioning protocol as per standard of care at the investigator's discretion followed by granulocyte colony-stimulating factor (GCSF)-mobilized human leukocyte antigen (HLA)-matched, related or unrelated donor allogeneic peripheral blood stem cells (unmanipulated), standard graft-versus-host disease (GVHD) prophylaxis as per standard of care at the investigator's discretion and rasburicase 0.20 mg/kg/day administered by intravenous infusion for 5 consecutive days. If after 5 days of rasburicase the participant's uric acid plasma level remains above 5 mg/dL, rasburicase may be continued for up to 7 days in total.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporin-A; Drug: etoposide; Drug: methotrexate; Drug: rasburicase; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation; Drug: fludarabine
- Control Group (Other): Historical chart review of patients from the Blood and Marrow Transplant database who received myeloablative allogeneic stem cell/bone marrow transplantation followed by standard GVHD prophylaxis in the past 10 years. Participants received allopurinol per institutional guidelines.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporin-A; Drug: etoposide; Drug: methotrexate; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation; Drug: fludarabine; Drug: allopurinol

INTERVENTIONS:
Drug: busulfan — Busulfan 3.2 mg/kg/day from day -7 to day -4 as standard of care for myeloablative (bone marrow depletion) conditioning at the investigator's discretion
Drug: cyclophosphamide — Cyclophosphamide as standard of care for myeloablative conditioning at the investigator's discretion
Drug: cyclosporin-A — Cyclosporin-A as standard of care for GVHD prophylaxis at the investigator's discretion
Drug: etoposide — Etoposide as standard of care for myeloablative conditioning at the investigator's discretion
Drug: methotrexate — Methotrexate 1.5 mg/kg/day on days -3, -2, and -1 as standard of care for GVHD prophylaxis at the investigator's discretion
Drug: rasburicase — Rasburicase 0.20 mg/kg intravenous infusion over 30 minutes for 5 to 7 days
  Arms: Rasburicase Group
Drug: sirolimus — Sirolimus as standard of care for GVHD prophylaxis at the investigator's discretion
Drug: tacrolimus — Tacrolimus as standard of care for GVHD prophylaxis at the investigator's discretion
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation — Total body irradiation 13.2 Gy over 8 fractions from day -7 to day - 4 for myeloablative conditioning at the investigator's discretion
Drug: fludarabine — Fludarabine 40 mg/m^2/day from day -6 to day -3 as myeloablative conditioning at the investigator's discretion
Drug: allopurinol — Allopurinol per institutional guidelines
  Arms: Control Group

SUMMARY:
RATIONALE: Rasburicase may be an effective treatment for graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This clinical trial is studying how well rasburicase works in preventing graft-versus-host disease in patients with hematologic cancer or other disease undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the incidence and severity of acute graft-vs-host disease (GVHD) in rasburicase-treated patients who will undergo myeloablative human leukocyte antigen (HLA)-matched related or unrelated donor allogeneic peripheral blood hematopoietic stem cell transplantation (SCT) for hematologic malignancies and compare these outcomes with those of historical controls.

Secondary

* To evaluate the efficacy (in terms of reduction of uric acid levels) and safety of rasburicase in patients undergoing myeloablative allogeneic SCT.
* To evaluate the graft-versus-host and host-versus-graft immune responses in rasburicase-treated patients.

OUTLINE: This is a multicenter study.

Patients receive a conventional myeloablative conditioning regimen consisting of high doses of cyclophosphamide, busulfan, and etoposide, with or without total-body irradiation. Depending on the preparative regimen selected, the conditioning of recipients will take a total of 6 to 7 days. On day 0, patients will receive filgrastim (G-CSF)-mobilized HLA-matched, related, or unrelated donor allogeneic peripheral blood stem cells (unmanipulated). Patients will receive standard graft-vs-host disease prophylaxis consisting of cyclosporine or tacrolimus and methotrexate or sirolimus. Patients will receive rasburicase IV over 30 minutes, beginning on the first day of conditioning therapy, for 5 consecutive days. If after 5 days of rasburicase the patient's uric acid plasma level remains above 5 mg/dL, rasburicase may be continued for up to 7 days in total.

Blood is obtained on day 0 and then at 14, 28, and 42 days post-transplant for immunologic studies, including quantitative analysis to follow the recovery of T cells, B cells, natural killer cells, dendritic cells (DC), and monocytes using flow cytometry (FCM); phenotypic analysis of T cells, DC and monocytes by FCM; lymphocyte activation analysis: CD3, CD4, CD8, CD25 2. CD3, CD8, CD71, CD69; DC analysis: CD45, CD14, DR, CD86, CD80 2. CD45, CD14, CD40, CD11c; and in vitro functional studies such as mixed lymphocyte reaction (MLR) and cell-mediated lysis (CML) to assess for the graft-versus-host and host-versus-graft responses. Peripheral blood is collected for chimerism studies on days 28 and 100 post-transplant.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with hematologic malignancies for whom conventional myeloablative allogeneic stem cell transplantation is deemed clinically appropriate and who are eligible for conventional myeloablative allogeneic stem cell transplantation on treatment plans/protocols, including any of the following:

  * Non-Hodgkin lymphoma or Hodgkin lymphoma (relapsed or refractory disease)
  * Chronic lymphocytic leukemia (received more than one previous treatment regimen)
  * Acute myelogenous or lymphoblastic leukemia (AML/ALL) (high-risk disease, in first complete remission [CR1] or subsequent remission, or primary refractory disease)
  * Chronic myelogenous leukemia in tyrosine-kinase resistant chronic phase, accelerated or blast phase, or primary refractory disease
  * Myelodysplastic syndromes in International Prognostic Scoring System (IPSS) high-intermediate or high-risk groups
  * Other hematologic disorders for which allogeneic stem cell transplantation is appropriate (e.g., myelofibrosis)
* Patients who have relapsed after standard autologous and/or allogeneic bone marrow transplant are eligible
* Must be receiving filgrastim (G-CSF)-mobilized related or unrelated donor allogeneic peripheral blood stem cells

  * Patients receiving hematopoietic stem cells of any other sources such as a marrow graft or umbilical cord blood will not be eligible for this study
* Donor must be HLA-genotypically or phenotypically 6 of 6 antigen matched (at the A, B, DR loci) related or unrelated

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Patients with a "currently active" second malignancy other than non-melanoma skin cancers can only be registered if survival from the second malignancy is expected to be more than 1 year
* Ejection fraction ≥ 45% by either radioisotope Multiple Gated Acquisition Scan (MUGA) scan or Echocardiogram (ECHO)
* Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) ≥ 50% of predicted with no symptomatic pulmonary disease
* Mini Mental Status Exam Score ≥ 20
* Patients must have an expected life expectancy of at least 3 months
* Patients with symptomatic visceral, blood stream or nervous system opportunistic infection are eligible if the infection has been appropriately treated and controlled

  * Patients with a fungal infection must have had treatment for at least one month and must have proof of regression of the infection prior to enrollment
  * Patients may be on antibiotics at the time of transplant

Exclusion criteria:

* Human Immunodeficiency Virus (HIV) infection
* Uncontrolled diabetes mellitus
* Active congestive heart failure from any cause

  * Previous history of congestive heart failure allowed
* Active angina pectoris
* Oxygen-dependent obstructive pulmonary disease
* Failure to demonstrate adequate compliance with medical therapy and follow-up
* Known history of Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency or history of hemolysis indicative of G6PD deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2013-02-12 (Actual); Study Completion 2013-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bimalangshu R. Dey, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yeh AC, Brunner AM, Spitzer TR, Chen YB, Coughlin E, McAfee S, Ballen K, Attar E, Caron M, Preffer FI, Yeap BY, Dey BR. Phase I study of urate oxidase in the reduction of acute graft-versus-host disease after myeloablative allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2014 May;20(5):730-4. doi: 10.1016/j.bbmt.2014.02.003. Epub 2014 Feb 12. PMID 24530972

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rasburicase Group | Control Group
Started | 25 | 21
Received Rasburicase Per Protocol | 24 | 0
Completed | 18 | 12
Not Completed | 7 | 9
Not completed — Death | 6 | 9
Not completed — Participant Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat participants included in the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasburicase Group | Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Full Range); unit: years] | 42.9 [20 to 59] | 45 [21 to 55] | 44 [20 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 14 | 9 | 23
Graft-Versus-Host Disease (GVHD) Prophylaxis Intervention [Count of Participants; unit: Participants] — Participants received GVHD prophylaxis at the investigator's discretion. MRD=matched related donor. MUD=matched unrelated donor. ATG=antithymocyte globulin.
  Participants
    MRD: Cyclsporine + Methotrexate | 14 | 11 | 25
    MRD: Tacrolimus + Methotrexate | 2 | 2 | 4
    MUD: Tacrolimus + Methotrexate + ATG | 4 | 8 | 12
    MUD: Tacrolimus + Methotrexate | 1 | 2 | 3
Conditioning Protocol Interventions [Count of Participants; unit: Participants]
  Busulfan + Cyclophosphamide | 12 | 16 | 28
  Busulfan + Fludarabine | 2 | 0 | 2
  Total Body Irradiation + Cyclophosphamide | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grades II to IV Acute Graft-Versus-Host Disease (aGVHD)
Description: aGVHD severity was determined using International Bone Marrow Transplant Registry (IBMTR) scale stage and grade of the skin, liver and gut. Stage 1: Skin=maculopapular rash <25% of body surface; Liver=Bilirubin 2-3 mg/dL and Gut=500-999 mL diarrhea/day or peristent nausea with histologic evidence of GvHD. Stage 2: Skin=maculopapular rash 25-50% of body surface; Liver=Bilirubin 3.1-6 mg/dL and Gut=1000-1499 mL diarrhea/day. Stage 3: Skin=maculopapular rash >50% of body surface; Liver=Bilirubin 6.1-15 mg/dL and Gut=≥1500 mL diarrhea/day. Stage 4: Skin=generalized erythroderma with bulla formation; Liver=Bilirubin >15 mg/dL and Gut=severe abdominal pain.
  Grade 1: Stage 1-2 rash; no liver or gut involvement. Grade II: Stage 3 rash, or stage 1 liver involvement, or stage 1 gut involvement. Grade III: None to stage 3 skin rash with stage 2-3 liver, or stage 2-4 gut involvement. Grade IV: Stage 4 skin rash, or stage 4 liver involvement.
Time Frame: Up to 71 months
Population: Intent-to-treat participants included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Rasburicase Group | Control Group
Number analyzed (Participants) | 21 | 21
percentage of participants | 24 | 57
Statistical Analysis 1: Comparison: Rasburicase Group vs Control Group; Test type: Superiority; p = .036, Gray's test for competing risks

2. Secondary Outcome: Uric Acid Levels
Description: Blood was collected and analyzed at a laboratory for serum uric acid levels reported in milligrams(mg)/deciliter(dL). Data is presented for those participants who experienced Grade II to IV aGVHD and those participants who did not experience Grade II to IV aGVHD at pre-transplant and post-transplant.
Time Frame: Pre-transplant Day -7 to Day -1 and Post-transplant Day 0 to Day 6
Population: Intent-to-treat population with data available for analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rasburicase Group | Control Group
Number analyzed (Participants) | 21 | 21
mg/dL
  Day -7 | 0.1 (0.209) | 4.157 (1.886)
  Day -6 | 0.075 (0.199) | 3.419 (1.752)
  Day -5 | 0.086 (0.24) | 2.967 (1.437)
  Day -4 | 0.1 (0.324) | 2.579 (1.249)
  Day -3 | 0.067 (0.2) | 2.358 (1.21)
  Day -2 | 0.081 (0.15) | 1.867 (1.097)
  Day -1 | 0.438 (0.611) | 1.71 (0.931)
  Day 0 | 0.938 (0.887) | 2.163 (1.012)
  Day 1 | 1.624 (1.205) | 2.671 (1.056)
  Day 2 | 2.076 (1.37) | 2.778 (0.985)
  Day 3 | 2.271 (1.303) | 2.805 (1.028)
  Day 4 | 2.548 (1.454) | 2.758 (1.161)
  Day 5 | 2.595 (1.729) | 2.579 (1.318)
  Day 6 | 2.705 (1.665) | 2.653 (1.33)

3. Secondary Outcome: Number of Participant With Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 71 months
Population: Safety population included all participants who received at least one dose of protocol specified treatment and were in remission at the time of transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Rasburicase Group | Control Group
Number analyzed (Participants) | 21 | 21
Participants | 21 | 21

4. Secondary Outcome: Graft-versus-host and Host-versus-graft Immune Responses
Description: Laboratory tests such as limited dilution assay (LDA) were to be performed to assess graft-versus-host and host-versus-graft immune responses.
Time Frame: Days -2, 0, and Days 14, 21 and 35 days post-transplant
Population: Due to laboratory and budgetary issues the planned laboratory testing and assays were not performed and no data were collected.
Arm/Group | Rasburicase Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 71 months
Description: Safety population included all participants who received at least one dose of protocol specified treatment and were in remission at the time of transplant.
Arm/Group | Rasburicase Group | Control Group
Serious Adverse Events (participants affected / at risk) | 10/21 | 9/21
Other Adverse Events (participants affected / at risk) | 21/21 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rasburicase Group (N=21) | Control Group (N=21)
Seizure (Nervous system disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Engraftment syndrome (Immune system disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 1 | 0
Relapsed disease (Blood and lymphatic system disorders) | 7 | 7 — Resulted in death
Infection from aGVHD flare (Infections and infestations) | 0 | 1 — Resulted in death
Respiratory failure (Infections and infestations) | 0 | 1 — Resulted in death
H1N1 influenza (Infections and infestations) | 1 | 0 — Resulted in death
Metapneumovirus (Infections and infestations) | 1 | 0 — Resulted in death
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rasburicase Group (N=21) | Control Group (N=21)
Vomiting (Gastrointestinal disorders) | 13 | 11
Fever (General disorders) | 5 | 9
Nausea (Gastrointestinal disorders) | 19 | 19
Diarrhea (Gastrointestinal disorders) | 15 | 9
Mucositis (General disorders) | 20 | 17
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Edema (Metabolism and nutrition disorders) | 5 | 2
Tongue numbness (Gastrointestinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes